CLINICAL TRIAL: NCT00000833
Title: A Phase I Study of Combination Therapy With Didanosine (ddI) and Ribavirin in HIV-Infected Children.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 274; 11250 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Ribavirin; Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Ribavirin; Didanosine

INTERVENTIONS:
Drug: Ribavirin
Drug: Didanosine

SUMMARY:
To compare the safety, toxicity, and tolerance of two doses of ribavirin in combination with didanosine (ddI) to HIV-infected children. To determine the toxicity of ddI/ribavirin and compare it to the expected toxicity of ddI monotherapy. To determine the effect of concurrent ribavirin on the pharmacokinetics of ddI. To determine a dosage of ribavirin that would be suitable for a Phase II/III evaluation of ddI/ribavirin.

Ribavirin, a broad spectrum antiviral agent, may enhance the antiretroviral activity of didanosine ( ddI ) without a concomitant increase in toxicity. Ribavirin alters the intracellular metabolism of ddI, enhancing the antiretroviral activity of the active form of ddI.

DETAILED DESCRIPTION:
Ribavirin, a broad spectrum antiviral agent, may enhance the antiretroviral activity of didanosine ( ddI ) without a concomitant increase in toxicity. Ribavirin alters the intracellular metabolism of ddI, enhancing the antiretroviral activity of the active form of ddI.

Patients are divided into two cohorts. Subjects will be stratified by age 3 months to < 24 months and >= 24 months to 12 years. Fifty % of patients from each age group will be assigned to each cohort. Cohort 1 receives ddI monotherapy for 4 weeks, followed by combination ddl/ribavirin therapy for an additional 20 weeks. Cohort 2 receives combination ddI/ribavirin for 24 weeks. In both cohorts, after study medications are stopped, patients are treated with prescription antiretrovirals for 4 more weeks. [AS PER AMENDMENT 7/2/96: Note: In each cohort of 10 subjects at least 2 of 5 children from the older half of the cohort will have an ICD p24 antigen at entry.]

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* Acetaminophen for no more than 72 hours.
* Immunoglobulin.
* Corticosteroids.
* Erythropoietin.
* G-CSF and GM-CSF.
* Ethionamide or isoniazid for TB if no alternative available.
* Immunizations according to current recommendations.

Patients must have:

* HIV infection.
* Immunologic abnormality or clinical symptoms as detailed in the Disease Status field.
* No active AIDS-defining opportunistic infection or malignancy, no progressive encephalopathy attributable to HIV and no chronic persistent diarrhea.
* Consent of parent or guardian.

PER AMENDMENT 7/2/96:

* At least 2 of the 5 children in the older half of each cohort must have an ICD p24 antigen concentration >= 70 pg/ml at screening.

Prior Medication:

Allowed:

* Up to 6 weeks of prior immunomodulator therapy.
* Maternal immunomodulator or antiretroviral therapy, including during pregnancy.
* Prior corticosteroids or intravenous immunoglobulin.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current grade 3 or worse neuropathy/lower motor neuropathy.
* Clinical or laboratory grade 3 or worse toxicities.
* Active serious bacterial infection.

Concurrent Medication:

Excluded:

* Chemotherapy for active malignancy.
* Antiretrovirals other than study drugs.
* Immunomodulators unless specifically allowed.

Patients with the following prior condition are excluded:

* History of grade 3 or worse neuropathy/lower motor neuropathy.

Prior Medication:

Excluded:

* Prior ddI or oral ribavirin.
* Aerosolized ribavirin within 6 weeks prior to study entry.
* Antiretroviral or immunomodulator therapy (other than corticosteroids or IVIG) within 1 week prior to blood draws for study entry.

Ongoing drug or alcohol abuse.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Van Dyke R, Study Chair; McSherry G, Study Chair
Locations (15):
- United States (14):
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Children's Hosp of Boston, Boston, Massachusetts
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp of New Jersey / UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Schneider Children's Hosp, New Hyde Park, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Glaxo Wellcome Inc, Research Triangle Park, North Carolina
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
- Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan, Puerto Rico

REFERENCES:
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173